CLINICAL TRIAL: NCT05844657
Title: Investigation of the Physical and Psychosocial Status and Quality of Life of People With Meniere's Disease
Brief Title: Comprehensive Evaluation in Patients With Meniere's Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gülistan Örenç, Physiotherapist (Student in Graduate School of Health Sciences), Hacettepe University
Other Study IDs: Hacettepe Universitey
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Meniere Disease; Psychosocial Problem; Physical Disability; Quality of Life
Keywords: Meniere's disease; postural balance; posture; vertigo; tinnitus; proprioception; quality of life
MeSH Terms: conditions — Meniere Disease; Vertigo; Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Meniere's disease: Voluntary Meniere's patients aged 18-65 years, not in the relapse period, who met the inclusion criteria
  Interventions: Other: Case report form; Other: Tinnitus disability scale; Other: A feeling of fullness and/or pressure in the ear; Other: Dizziness intensity and frequency; Other: Dizziness disability inventory; Other: Vertigo symptom scale-short form; Other: Hearing Impairment Scale; Other: Cervical Range of Motion (CROM 3) device; Other: Temporomandibular joint range of motion assessment; Other: Posture evaluation with New York posture analysis; Other: Evaluation of the anterior tilt angle of the head; Other: Evaluation of postural balance with the Freemed pressure platform; Other: Static balance assessment with tandem stance test; Other: Dynamic balance assessment with tandem gait test; Other: Headache, Temporomandibular pain and Craniocervical pain presence and severity assessment; Other: Pain sensitivity assessment in the head, neck, shoulder girdle and upper back region; Other: International physical activity questionnaire-measurement of physical activity level with short; Other: Evaluation of sleep quality with the Pittsburgh sleep quality index; Other: Evaluation of fatigue with the fatigue severity scale; Other: Evaluation of anxiety-depression status with hospital anxiety and depression scale; Other: Evaluation of quality of life with short form-12 (SF-12); Other: the International Fall Efficiency Scale; Other: assessment of muscle performance
- Healthy individuals without Meniere's disease: Volunteer healthy individuals aged 18-65 years without dizziness who met the inclusion criteria
  Interventions: Other: Case report form; Other: Tinnitus disability scale; Other: A feeling of fullness and/or pressure in the ear; Other: Dizziness intensity and frequency; Other: Dizziness disability inventory; Other: Vertigo symptom scale-short form; Other: Hearing Impairment Scale; Other: Cervical Range of Motion (CROM 3) device; Other: Temporomandibular joint range of motion assessment; Other: Posture evaluation with New York posture analysis; Other: Evaluation of the anterior tilt angle of the head; Other: Evaluation of postural balance with the Freemed pressure platform; Other: Static balance assessment with tandem stance test; Other: Dynamic balance assessment with tandem gait test; Other: Headache, Temporomandibular pain and Craniocervical pain presence and severity assessment; Other: Pain sensitivity assessment in the head, neck, shoulder girdle and upper back region; Other: International physical activity questionnaire-measurement of physical activity level with short; Other: Evaluation of sleep quality with the Pittsburgh sleep quality index; Other: Evaluation of fatigue with the fatigue severity scale; Other: Evaluation of anxiety-depression status with hospital anxiety and depression scale; Other: Evaluation of quality of life with short form-12 (SF-12); Other: the International Fall Efficiency Scale; Other: assessment of muscle performance

INTERVENTIONS:
Other: Case report form — Sociodemographic information (age, gender, height, body mass index, marital status, occupation, education level, contact information), frequency of smoking and alcohol use, frequency of caffeine consumption, frequency of salt consumption, dominant side, background, family history, medical and audiological information were recorded.
Other: Tinnitus disability scale — Tinnitus disability scale was used to evaluate the tinnitus severity of Meniere's patients. It consists of 25 items in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'. Tinnitus level or severity is determined by calculating the total score of the answers given.
Other: A feeling of fullness and/or pressure in the ear — The feeling of fullness or pressure in the ear was evaluated verbally by receiving yes/no responses from the participants.
Other: Dizziness intensity and frequency — In order to determine the frequency and severity of dizziness, the participants were asked to mark the appropriate score between 1-10 points.
Other: Dizziness disability inventory — The dizziness disability inventory was used to determine the disability level of the individuals participating in our study. It consists of 25 questions in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'.
Other: Vertigo symptom scale-short form — The short form of the vertigo symptom scale was used to determine the frequency and duration of vertigo in the individuals participating in our study. The vertigo symptom scale consisting of 8 questions consists of vertigo (VSS-V), and the vertigo symptom scale consisting of 7 questions consists of two subsections consisting of a total of 15 questions: anxiety (VSS-A). Each item; Never (0), Very rarely (1 point), Often (2 points), Often - every week (3 points), Very often - On average, at least twice a week (4 points). The total score ranges from 0 to 60.
Other: Hearing Impairment Scale — The Adult Hearing Impairment Scale was used to determine the effect of the current hearing impairment levels of the individuals participating in our study on their daily living activities. The scale consists of 25 questions in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'. Participants mark the most appropriate expression for them.
Other: Cervical Range of Motion (CROM 3) device — "Cervical Range of Motion" (CROM) device was used to evaluate the sense of proprioception and range of motion (ROM) in the cervical region muscles. A total of six positions were performed: right cervical rotation, left cervical rotation, right cervical lateral flexion, left cervical lateral flexion, cervical extension and cervical flexion.
Other: Temporomandibular joint range of motion assessment — In our study, the temporamandibular joint range of motion (ROM) was evaluated with a ruler specific to each participant in four positions, including mandibular depression, protraction, and right and left lateral deviation.
Other: Posture evaluation with New York posture analysis — The New York Posture Evaluation method was used to obtain information about the general posture correctness of the participants. Posture changes that may occur in 13 different parts of the body, 7 from the side and 6 from the back, including the head, neck, shoulder, back, waist, hip and ankle, were examined in the anatomical position of the individuals. As a result of the observation, the posture of the individual was scored according to whether it was severely bad (1 point), moderately bad (3 points), and straight (5 points). The total score obtained varies between 13-65.
Other: Evaluation of the anterior tilt angle of the head — Anterior tilt angles of the head of the participants were evaluated with photographs taken from the lateral (lateral) side. The anterior tilt angle was calculated as the angle between the line drawn between the C7 cervical spinous process and the tragus and the straight line drawn vertically from C7.
Other: Evaluation of postural balance with the Freemed pressure platform — Postural sway and lower extremity weight transfer were evaluated with the Freemed baropodometric pressure platform (Rome, Italy) system, which has been shown to be valid and reliable.
Other: Static balance assessment with tandem stance test — In our study, the tandem stance test was used for static evaluation. A total of four assessments were made on the participants, first with their right foot in front, eyes open and eyes closed, then left foot in front with eyes open and eyes closed.
Other: Dynamic balance assessment with tandem gait test — In our study, the tandem gait test was used for dynamic evaluation. A straight line was created with a white tape attached to the floor, almost 2 feet away from the 10-foot-long wall. The participant was asked to walk along the line created by taping the heel of the forward foot to touch the toe of the back foot, at a comfortable pace in daily life and with eyes open.
Other: Headache, Temporomandibular pain and Craniocervical pain presence and severity assessment — Headache, temporomandibular pain and craniocervical pain were asked to mark the person from the photographs taken from the front, back and side in the form of a human figure. Pain severity was evaluated with the numerical rating scale (NRS).
Other: Pain sensitivity assessment in the head, neck, shoulder girdle and upper back region — In our study, muscle tenderness was evaluated by manual pressure algometry and palpation. Muscle tenderness was assessed in the upper and lower regions of the masseter, temporalis, sternocleidomastoid, and upper trapezius muscles on both right and left sides.
Other: International physical activity questionnaire-measurement of physical activity level with short — The short form of the international physical activity questionnaire was used to determine the physical activity level of the individuals participating in our study. The short form of the international physical activity questionnaire evaluates the last week and consists of a total of 4 sections and 7 questions. Duration of physical activity that requires intense physical effort, such as heavy lifting, soccer, or fast cycling; times of doing moderate physical activities that cause breathing slightly more often than usual; The total duration of walks at work, home, for sports, exercise and hobby, and the total sitting time spent in a day at work, at home or while resting are calculated.
Other: Evaluation of sleep quality with the Pittsburgh sleep quality index — The Pittsburgh Sleep Quality Index (PUKI) was used to evaluate the sleep quality and disturbance of the individuals participating in our study in the last month. It consists of a total of 24 questions. The participant responds to each item according to the frequency between 0-3 points. The total score (0-21 points) from these components indicates whether the sleep quality is good or not.
Other: Evaluation of fatigue with the fatigue severity scale — The Fatigue severity scale was used to evaluate the fatigue status of the individuals participating in our study. The scale uses a scoring system ranging from 1-7, which starts as I do not agree (1 point) and increases gradually towards I agree (7 point). It consists of 9 items in total and people mark the option that suits them.
Other: Evaluation of anxiety-depression status with hospital anxiety and depression scale — The Hospital Anxiety and Depression Scale (HADS) was used to evaluate the anxiety and depression status of the individuals participating in our study. For each item, the participant answers with a four-point (0-3 points) response option. Therefore, the possible score probabilities in line with the answers given are minimum '0' and maximum '21'. The cut-off point for the anxiety subscale is 10 points, while the cut-off point for the depression subscale is 7 points.
Other: Evaluation of quality of life with short form-12 (SF-12) — The Short form SF-12 Questionnaire was used to evaluate the quality of life of the individuals participating in our study. The summary score of the physical and mental components varies between 0-100, and the higher the score in the components, the better the quality of life.
Other: the International Fall Efficiency Scale — The International Fall Activity Scale (UDES) was used to evaluate both the attack and the general fear of falling of the individuals participating in our study. It consists of 16 questions in total. The answer to each question is marked on a scale between 1 and 4 points. Expressions such as I never worry (1 point), I worry a little (2 point), I am very worried (3 point), I am very worried (4 point) are used as the level of anxiety increases as the score increases. The total score obtained ranges from 16 (no worries) to 64 (extremely worried).
Other: assessment of muscle performance — In our study, the strength of cervical flexors, anterior and oblique trunk flexors, cervical extensor muscles, back extensor muscles, trapezius muscle, and rhomboid major-minor muscles were evaluated. In addition, the endurance of the deep cervical flexor muscles, cervical flexors and cervical extensor muscles were also evaluated.

SUMMARY:
The aim of our study is to determine the severity of the disease in people with Meniere's Disease; physical conditions such as balance, posture, pain, physical activity level, neck joint range of motion, proprioception; to examine psychosocial conditions such as depression, anxiety, sleep quality, fatigue, and quality of life and to make a comprehensive evaluation by comparing it with healthy volunteers.

DETAILED DESCRIPTION:
Meniere's disease (MD) is an inner ear disease characterized by independent attacks and lasting for at least 20 minutes, dizziness, recurrent hearing loss during seizures, tinnitus, fullness in the ear, and a feeling of headache. After the diagnosis of the disease, the most disturbing situation for the patient is the uncertainty of the progression of the disease and the deterioration of the quality of life. It is very difficult to know and predict how the disease will progress. Quality of life is impaired by current symptoms and may be further reduced by uncertainty about when another attack may occur and activity restriction due to fear of provoking symptoms with exertion or stress.

When the studies on MD are examined, it is seen that the symptoms affect not only certain physical conditions but also psychological conditions. It has been observed that psychological factors play a more important role than is commonly realized in terms of their impact on patients' quality of life. MD has a negative impact on the person's daily life, and the person avoids certain daily activities or situations because of the illness. Looking at the literature, it is not known whether the severity of disease symptoms or whether the psychological state precedes the physical state.

In light of all this information, MD appears to be a multifaceted condition that can have major and often alarming effects on the lives of affected individuals. Therefore, it is important to evaluate individuals with MD with a holistic approach.

The aim of our study is to determine the severity of the disease in people with Meniere's Disease; physical conditions such as balance, posture, pain, physical activity level, neck joint range of motion, proprioception; to examine psychosocial conditions such as depression, anxiety, sleep quality, fatigue, and quality of life and to make a comprehensive evaluation by comparing it with healthy volunteers.

ELIGIBILITY:
Study group Inclusion Criteria:

* Having been diagnosed with Meniere's disease as a result of clinical and audiological evaluation by an ENT specialist
* ability to read and write
* be between the ages of 18-65
* Not having an acute attack and not receiving acute attack treatment during the study period,
* Having given consent to participate in the study as a result of the information
* A minimum score of 24 on the Mini Mental Test (MMDT)

Study group Exclusion Criteria:

* Known neurological disease (head trauma, spinal trauma, multiple sclerosis, intracranial tumor, etc.) Having an anatomical problem or disease related to the outer and middle ear
* Peripheral and central vestibular pathology other than Meniere's disease
* Sensorineural hearing loss due to other causes
* Other neurological, orthopedic, circulatory system or vision problems that may cause vertigo, dizziness and balance disorder

Control group Inclusion Criteria:

* ability to read and write
* be between the ages of 18-65
* Not having an acute attack and not receiving acute attack treatment during the study period,
* Having given consent to participate in the study as a result of the information
* A minimum score of 24 on the Mini Mental Test (MMDT)
* without vertigo

Control group Exclusion Criteria:

* suffering from vertigo
* Known neurological disease (head trauma, spinal trauma, multiple sclerosis, intracranial tumor, etc.) Having an anatomical problem or disease related to the outer and middle ear
* Peripheral and central vestibular pathology other than Meniere's disease
* Sensorineural hearing loss due to other causes
* Other neurological, orthopedic, circulatory system or vision problems that may cause vertigo, dizziness and balance disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with Meniere's disease and people with without Meniere's disease
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Evaluating the sense of proprioception with the "Cervical Range of Motion" (CROM) device | March 2023- May 2023
  "Cervical Range of Motion" (CROM) device was used to evaluate the sense of proprioception. A total of six positions were performed: right cervical rotation, left cervical rotation, right cervical lateral flexion, left cervical lateral flexion, cervical extension and cervical flexion.
Evaluation of the range of motion (ROM) in the cervical region muscles with the "Cervical Range of Motion" (CROM) device | March 2023-May 2023
  "Cervical Range of Motion" (CROM) device was used to evaluate the range of motion (ROM) in the cervical region muscles. A total of six positions were performed: right cervical rotation, left cervical rotation, right cervical lateral flexion, left cervical lateral flexion, cervical extension and cervical flexion.
Temporomandibular joint range of motion assessment | March 2023- May 2023
  In our study, the temporamandibular joint range of motion (ROM) was evaluated with a ruler specific to each participant in four positions, including mandibular depression, protraction, and right and left lateral deviation.
Posture evaluation with New York posture analysis | March 2023- May 2023
  The New York Posture Evaluation method was used to obtain information about the general posture correctness of the participants. Posture changes that may occur in 13 different parts of the body, 7 from the side and 6 from the back, including the head, neck, shoulder, back, waist, hip and ankle, were examined in the anatomical position of the individuals. As a result of the observation, the posture of the individual was scored according to whether it was severely bad (1 point), moderately bad (3 points), and straight (5 points). The total score obtained varies between 13-65.
Evaluation of the anterior tilt angle of the head | March 2023- May 2023
  Anterior tilt angles of the head of the participants were evaluated with photographs taken from the lateral (lateral) side. The anterior tilt angle was calculated as the angle between the line drawn between the C7 cervical spinous process and the tragus and the straight line drawn vertically from C7.
Evaluation of postural balance with the Freemed pressure platform | March 2023- May 2023
  Postural sway and lower extremity weight transfer were evaluated with the Freemed baropodometric pressure platform (Rome, Italy) system, which has been shown to be valid and reliable.
Static balance assessment with tandem stance test | March 2023- May 2023
  In our study, the tandem stance test was used for static evaluation. A total of four assessments were made on the participants, first with their right foot in front, eyes open and eyes closed, then left foot in front with eyes open and eyes closed.
Dynamic balance assessment with tandem gait test | March 2023- May 2023
  In our study, the tandem gait test was used for dynamic evaluation. A straight line was created with a white tape attached to the floor, almost 2 feet away from the 10-foot-long wall. The participant was asked to walk along the line created by taping the heel of the forward foot to touch the toe of the back foot, at a comfortable pace in daily life and with eyes open.
Headache presence and severity assessment | March 2023- May 2023
  The participant was asked to mark the places where the headache occurred from the photographs taken in the form of a human figure from the front, back and side. Pain severity was evaluated with the Numerical Rating Scale. The lowest score 0 indicates 'I have no pain' and the highest score 10 indicates 'I have unbearable pain'. As the score increases, the severity of pain increases.
Craniocervical pain presence and severity assessment | March 2023-May 2023
  The participant was asked to mark the areas of craniocervical pain from the photographs taken in the form of a human figure from the front, back and side. Pain severity was evaluated with the Numerical Rating Scale. The lowest score 0 indicates 'I have no pain' and the highest score 10 indicates 'I have unbearable pain'. As the score increases, the severity of pain increases.
Temporomandibular pain presence and severity assessment | March 2023-May 2023
  The participant was asked to mark the places where temporomandibular pain occurred from the photographs taken in the form of a human figure from the front, back and side. Pain severity was evaluated with the Numerical Rating Scale. The lowest score 0 indicates 'I have no pain' and the highest score 10 indicates 'I have unbearable pain'. As the score increases, the severity of pain increases.
Pain sensitivity assessment in the head, neck, shoulder girdle and upper back region | March 2023- May 2023
  In our study, muscle tenderness was evaluated by manual pressure algometry and palpation. Muscle tenderness was assessed in the upper and lower regions of the masseter, temporalis, sternocleidomastoid, and upper trapezius muscles on both right and left sides.
Evaluation of sleep quality with the Pittsburgh sleep quality index | March 2023- May 2023
  The Pittsburgh Sleep Quality Index was used to evaluate the sleep quality and discomfort of the individuals participating in our study in the last month. It consists of a total of 24 questions. The participant answers each item between 0-3 points according to the frequency. The total score (0-21 points) from these components indicates whether the sleep quality is good or not. As the total score increases, sleep quality decreases and sleep disorder status increases. A total score of 5 or more indicates poor sleep quality.
Evaluation of fatigue with the fatigue severity scale | March 2023- May 2023
  The Fatigue Severity Scale was used to evaluate the fatigue status of the individuals participating in our study. The Fatigue Severity Scale uses a scoring system ranging from 1-7, starting with disagree (1 point) and gradually increasing to agree (7 points). It consists of 9 items in total and people mark the option that suits them. Possibilities of total points that can be taken vary between 9-63 points. A score of 36 and above indicates that the level of fatigue is severe. The higher the score, the higher the level of fatigue.
Evaluation of anxiety-depression status with hospital anxiety and depression scale | March 2023- May 2023
  The Hospital Anxiety and Depression Scale was used to evaluate the anxiety and depression status of the individuals participating in our study. The participant answers with a four-point (0-3 point) response option for each item. Therefore, according to the answers given, the possible score probabilities are minimum '0' and maximum '21'. The cut-off point for the anxiety subscale is 10 points, and the cut-off point for the depression subscale is 7 points. The higher the total score, the higher the level of depression and anxiety.
Evaluation of quality of life with short form-12 (SF-12) | March 2023- May 2023
  The Short form SF-12 Questionnaire was used to evaluate the quality of life of the individuals participating in our study. The summary score of the physical and mental components varies between 0-100, and the higher the score in the components, the better the quality of life.
the International Fall Efficiency Scale | March 2023- May 2023
  The International Fall Activity Scale (UDES) was used to evaluate both the attack and the general fear of falling of the individuals participating in our study. It consists of 16 questions in total. The answer to each question is marked on a scale between 1 and 4 points. Expressions such as I never worry (1 point), I worry a little (2 point), I am very worried (3 point), I am very worried (4 point) are used as the level of anxiety increases as the score increases. The total score obtained ranges from 16 to 64.

SECONDARY OUTCOMES:
Tinnitus disability scale | March 2023- May 2023
  Tinnitus disability scale was used to evaluate the tinnitus severity of Meniere's patients. It consists of 25 items in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'. Tinnitus level or severity is determined by calculating the total score of the answers given.
A feeling of fullness and/or pressure in the ear | March 2023- May 2023
  The feeling of fullness or pressure in the ear was evaluated verbally by receiving yes/no responses from the participants.
Dizziness intensity and frequency | March 2023- May 2023
  In order to determine the frequency and severity of dizziness, the participants were asked to mark the appropriate score between 1-10 points. 1 point indicates no dizziness, 10 points indicates continuous and extremely severe dizziness. As the score increases, the frequency and severity of dizziness also increase.
Dizziness disability inventory | March 2023- May 2023
  The dizziness disability inventory was used to determine the disability level of the individuals participating in our study. It consists of 25 questions in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'.
Vertigo symptom scale-short form | March 2023- May 2023
  The short form of the vertigo symptom scale was used to determine the frequency and duration of vertigo in the individuals participating in our study. The vertigo symptom scale consisting of 8 questions consists of vertigo (VSS-V), and the vertigo symptom scale consisting of 7 questions consists of two subsections consisting of a total of 15 questions: anxiety (VSS-A). Each item; Never (0), Very rarely (1 point), Often (2 points), Often - every week (3 points), Very often - On average, at least twice a week (4 points). The total score ranges from 0 to 60.
Hearing Impairment Scale | March 2023- May 2023
  The Adult Hearing Impairment Scale was used to determine the effect of the current hearing impairment levels of the individuals participating in our study on their daily living activities. The scale consists of 25 questions in total. The questions are scored between 0-2-4. It is calculated as 'Yes (4 points)', 'Sometimes (2 points)', 'No (0 points)'. Participants mark the most appropriate expression for them.
International physical activity questionnaire-measurement of physical activity level with short | March 2023- May 2023
  The short form of the international physical activity questionnaire was used to determine the physical activity levels of the individuals participating in our study. The short form of the international physical activity questionnaire evaluates the last week and consists of a total of 4 sections and 7 questions. The duration of physical activity that requires intense physical exertion, such as heavy lifting, soccer, or fast cycling; times of doing moderate physical activities that cause breathing slightly more often than usual; The total duration of walks at work, home, sports, exercise and hobby, and the total sitting time spent in a day at work, at home or while resting are calculated. The physical activity score is calculated by converting the Metabolic Equivalent of Task, which corresponds to the basal metabolic rate. Total Metabolic Equivalent of Task value varies between 0-3000. The higher the total score, the higher the level of physical activity.
Assessment of muscle strength | March 2023- May 2023
  In our study, the strength of cervical flexors, anterior and oblique trunk flexors, cervical extensor muscles, back extensor muscles, trapezius muscle and rhomboid major-minor muscles were evaluated.
Evaluation of muscle endurance | March 2023- May 2023
  In our study, the endurance of deep cervical flexor muscles, neck cervical flexors and neck cervical extensor muscles were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nezire Kose, Study Director — Hacettepe University, Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe Sağlık Bilimleri Enatitüsü, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorne A, Agerberg G. Craniomandibular disorders in patients with Meniere's disease: a controlled study. J Orofac Pain. 1996 Winter;10(1):28-37. PMID 8995914
- [Background] Bjorne A, Agerberg G. Symptom relief after treatment of temporomandibular and cervical spine disorders in patients with Meniere's disease: a three-year follow-up. Cranio. 2003 Jan;21(1):50-60. doi: 10.1080/08869634.2003.11746232. PMID 12555932
- [Background] Yardley L, Dibb B, Osborne G. Factors associated with quality of life in Meniere's disease. Clin Otolaryngol Allied Sci. 2003 Oct;28(5):436-41. doi: 10.1046/j.1365-2273.2003.00740.x. PMID 12969347
- See also: Craniomandibular disorders in patients with Menière's disease: a controlled study — https://pubmed.ncbi.nlm.nih.gov/8995914/
- See also: Symptom relief after treatment of temporomandibular and cervical spine disorders in patients with Meniere's disease: a three-year follow-up — https://pubmed.ncbi.nlm.nih.gov/12555932/
- See also: Factors associated with quality of life in Menière's disease — https://pubmed.ncbi.nlm.nih.gov/12969347/